CLINICAL TRIAL: NCT03162640
Title: Link Between Impulsivity and Time Anticipation
Brief Title: Impulsivity and Time Perception
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6526
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2017-05

CONDITIONS: Cannabis Use
Keywords: Early onset of cannabis use; Addiction; Time perception
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- P: for cannabis
- C: for the control group

SUMMARY:
Cannabis smokers having begun prematurely their consumption (before 16 years) present a persistent impulsivity much later after have stopped their consumptions. The literature highlights that the impulsivity promotes the passage towards a compulsive consumption, and the loss of control. To explain this phenomenon, some authors hypothesized that impulsivity would lead the subjects to overestimate the duration of events and to choose immediate rewards than preferred but delayed rewards. This hypothesis questions the role of the temporal anticipation in the impulsive choices. In a first hypothesis, the temporal impulsivity could be an endogenous deficit bound to the reward, and would be responsible for disorders of the temporal anticipation. In this case, the disorders should be observed especially when the subject anticipates a reward. Alternately, a disorder of the temporal anticipation could provoke impulsivity, and in this case, would be present with or without reward. To separate these hypotheses, we propose to test the capacities of temporal anticipation of non-smokers and early smokers of cannabis by means of a behavioral task " Hazard function task ", which allow to measure the capacity of a subject to anticipate the apparition of an event on the basis of a temporal cue. The neuronal correlates will be measured by a recording EEG of the wave ' CNV ' (fix a quota for denial of variation) which reflects the temporal accumulation and the processes of anticipation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers Man or woman of age between 18 and 50 years-old
* Absence of consumption of cannabis and tobacco for 1 year and absence of substance use disorder in history
* Matching in age and sex to the group consumers of cannabis
* Early consumers of cannabis (at the beginning of the consumptions before 16 years)
* Man or woman of age between 18 and 50 years old
* Statement of more than three consumptions a day of cannabis for at least one year and consumption of cannabis having begun before the age of 16 years.
* Urinary analysis is positive for the presence of cannabis
* Positive auto-questionnaire CAST: 2 positive answers to CAST questionnaire
* Hospitalized or not

Exclusion Criteria:

* Presence or history of a severe and invalidating somatic pathology (neurological, cardiovascular, lung, metabolic, renal, hepatic, gastro-intestinal)

  * History of cranial trauma with loss of consciousness.
  * substance use disorder except the substance tested in the protocol (cannabis).
  * Invalidating sensory disorders in particular visual: glaucoma, any retinal pathology. Visual acuteness 0.8
  * History of general anesthesia in the previous 3 months the study
  * Any evolutionary neurological or psychiatric pathology
  * Subject under guardianship
  * pregnancy
  * Feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cannabis use Versus Non-smokers
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Measure the capacities of the subjects to anticipate the apparition of the target | 8 days after inclusion in the study
  on the basis of a temporal cue presented before the target, and give the response as quickly as possible after the presentation of a rewarding versus not rewarding target.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence LALANNE-TONGIO, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace, France

IPD SHARING:
Plan to Share IPD: No